CLINICAL TRIAL: NCT05169645
Title: STOP CSUA: phySical acTivity, mOod and sleeP in Chronic Spontaneous Urticaria and
Brief Title: STOP CSUA: phySical acTivity, mOod and sleeP in Chronic Spontaneous Urticaria and Angioedema
Acronym: STOP CSUA
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: St. James's Hospital, Ireland (Other)
Responsible Party: Principal Investigator, Dr. Katie Ridge, Immunology specialist registrar, St. James's Hospital, Ireland
Other Study IDs: ATHENACX
Record Dates: First submitted 2021-12-13; First posted 2021-12-27 (Actual); Last update posted 2021-12-27 (Actual); Status verified 2021-12

CONDITIONS: Chronic Spontaneous Urticaria
MeSH Terms: conditions — Chronic Urticaria

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CSUA patients: CSUA patients
  Interventions: Other: Physical activity monitoring - Symptom monitoring

INTERVENTIONS:
Other: Physical activity monitoring - Symptom monitoring — This is an observational study. There is no intervention outside the collection of data from participants. Consenting participants in the study will be provided with a Fitbit activity tracker and asked to wear it for a period of three months.
  The Fitbit measures:
  * Physical activity using daily step count
  * Additional physical activity entries
  * Heart rate
  * Sleep quality
  * Calories burned
  * Food log
  Participants will be asked to download an app onto their smart phone entitled Athena CX. This app is designed to capture:
  * Urticaria symptomatology using the urticaria control test
  * Symptoms of depression using 2 items from the PHQ 9
  * Symptoms of anxiety using two items from the GAD
  * Short form self-compassion scale

SUMMARY:
Chronic spontaneous urticaria and angioedema (CSUA) is a disease of the skin characterised by hives, swellings or both that last longer than 6 weeks. People with this disease commonly describe poor sleep, reduced quality of life and psychological difficulties such as depression and anxiety. This study seeks to understand relationships between physical activity, sleep and symptoms of urticaria. We are asking individuals with urticaria to wear a fitbit tracker which monitors their physical activity and sleep. Participants also download an app onto their smartphone called Athena CX which is designed by the study team in DCU. The purpose of the app is capture real-time information from participants on mood and any skin symptoms they experience. We will use this information to learn more about possible links between symptoms of urticaria and lifestyle behaviours.

DETAILED DESCRIPTION:
Chronic spontaneous urticaria and angioedema (CSUA) is a disease of the skin characterised by hives, swellings or both that last longer than 6 weeks (1). A quarter of patients with this disease report impaired quality of life (2). Furthermore, individuals with CSUA are more likely to have depression and anxiety (3). In addition, our previous qualitative research findings have noted issues with self-compassion among this cohort (4). Fatigue and poor sleep are common (5). We seek to examine possible links between physical activity, sleep, mood and symptoms of urticaria.

For participants who give their consent, we will do this by collecting and exploring:

* Fitbit tracker data
* Information on mood via the Athena CX app
* Information on symptoms of urticaria via the Athena CX app

Electronic health applications for smartphones are increasingly used in chronic health conditions and have been piloted in chronic spontaneous urticaria for recording of symptoms, medication reminders and patient education. This study will develop a smartphone application designed specifically for this cohort of patients, entitled Athena CX focusing specifically upon symptomatology and mood.

An observational study collecting biofeedback data in this cohort will inform our understanding of this disease and future research.

Objectives

1. To delineate the psychological symptoms encountered by this cohort of patients
2. To examine whether there is a link between biofeedback data and symptoms of chronic spontaneous urticaria and angioedema (CSUA)
3. To collect linked clinical data on participants with CSUA
4. To inform an RCT examining the use of a digital behavioural intervention for patients with CSUA

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of chronic spontaneous urticaria with or without angioedema
2. Urticaria control test score < 12 indicating poorly controlled urticaria at time of consent
3. Preference to participate in the study
4. In possession of a smartphone

Exclusion Criteria:

Unable or unwilling to provide informed consent

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Chronic spontaneous urticaria clinic
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2022-02-01 (Estimated); Primary Completion 2022-09-01 (Estimated); Study Completion 2023-02-01 (Estimated)

PRIMARY OUTCOMES:
Physical activity | Followed for 12 weeks during programme
  Step count as measured by fitbit
Urticaria symptomatology | Followed for 12 weeks during programme
  Urticaria control test score
Heart rate variability | Followed for 12 weeks during programme
  Heart rate variability

CONTACTS AND LOCATIONS:
Overall Officials: Niall Conlon, Principal Investigator — St. James's Hospital, Ireland
Locations (1):
- St. James's Hospital, Dublin, Ireland

IPD SHARING:
Plan to Share IPD: Undecided